CLINICAL TRIAL: NCT03284372
Title: Safer Food Allergy Management for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 827073
Record Dates: First submitted 2017-09-07; First posted 2017-09-15 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Food Allergy; Adherence, Medication
MeSH Terms: conditions — Food Hypersensitivity; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intervention 1 (Experimental): Text Message Only
  Interventions: Behavioral: Text Message Only
- Intervention 2, Incentive (Experimental): Text message + Incentive
  Interventions: Behavioral: Text message + Incentive 1
- Cohort (No Intervention): For the cohort multiple randomized controlled trial (cmRCT), investigators will recruit 130 participants (the base cohort) ages 15-19. The base cohort allows investigators to measure normative food allergy self-management practices, while also serving as a control for experiments in Interventions 1 and 2.
- Control (No Intervention): The baseline cohort serves as the control group in this cmRCT. Participants will not receive text message reminders (during Intervention 1) or incentives (during Intervention 2). However, they will participate in all data collection points, including text message check-ins to assess epinephrine-carrying. Participants in the base cohort will receive usual care.
- Adolescent Allergy Advisors (No Intervention): We will pilot the text messages to be used in Interventions 1 and 2 through interviews and cognitive testing among 20 Adolescent Allergy Advisors, who will critique message content, framing, and language. These advisors will not be part of the cohort multiple randomized controlled trial.

INTERVENTIONS:
Behavioral: Text Message Only — The intervention group (n=25, randomly selected from the base cohort) will receive informational and socially supportive text messages during a 10-week intervention. Investigators will deploy the intervention using the Way to Health platform, which automates outgoing messages and feedback. Many of the messages will be sent to all Intervention 1 participants, to assure consistency of the intervention. A subset will be tailored to address participants' specific allergies. At 10 unannounced check-ins, we will send text messages asking participants in the intervention and control groups if they are carrying their epinephrine.
  Arms: Intervention 1
Behavioral: Text message + Incentive 1 — Among base cohort members not exposed to the text message only intervention (#1), we will randomly select a new intervention group (n=50) to receive text message reminders plus Incentive 1. At each of 10 unannounced check-ins, if unsuccessful in documenting epinephrine-carrying, participants will lose part of their incentive. The remainder of the Cohort (control) will receive text reminders.
  Arms: Intervention 2, Incentive

SUMMARY:
Among the 15 million people with food allergies in the U.S., adolescents experience the highest risk of adverse events. Yet, there are few evidence-based strategies to improve food allergy management in adolescents. In a cohort multiple randomized controlled trial, this study will include two experiments to test the effectiveness of text message reminders and incentives to encourage epinephrine-carrying.

DETAILED DESCRIPTION:
Among the 15 million people with food allergies in the United States, adolescents experience the highest risk of adverse events, including death from anaphylaxis. Visits to one pediatric emergency department for anaphylaxis doubled between 2001 and 2006, suggesting a rapidly escalating public health burden. Despite this critical concern, there are few evidence-based strategies to improve food allergy management in adolescents, who must sustain three core prevention strategies: diligent avoidance of allergenic foods, consistent carrying of potentially life-saving epinephrine auto-injectors, and prompt administration of epinephrine in the event of anaphylaxis.

The objective of this study is to develop and test interventions to encourage safer food allergy management among adolescents. The primary outcome is consistency of epinephrine-carrying, measured using cell phone photographs at randomly-timed check-ins. This study will be among the first to longitudinally track normative food allergy management practices and one of the first to test behavior change strategies.

In a cohort multiple randomized controlled trial (n=130), the study will include two experiments to test the effectiveness of text message reminders and incentives, using various incentive designs that have proven effective in prior behavioral economics interventions to encourage weight loss and smoking cessation. Aim 1. Test the impact of a text-message reminder system on consistency of epinephrine carrying. Aim 2. Test the impact of modest incentives on consistency of epinephrine carrying. Based on promising preliminary data, the central hypothesis is that, compared to controls, adolescents who receive text message reminders plus modest financial incentives will more consistently carry their epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* Food allergy diagnosis by a physician and recorded in the medical chart
* Prior prescription of epinephrine auto-injector to treat anaphylaxis
* Access to a cell phone capable of sending and receiving text messages and photographs (our team will provide cell phones to participants willing to participate, but who do not own a cellphone)
* Fluent in English
* Between ages 15-19 at baseline

Exclusion Criteria:

* Unable to obtain permission (consent) of a parent to participate in the study
* Will not or cannot give assent
* Currently participating in another clinical trial with related aims

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of check-ins at which participant is carrying epinephrine auto-injector | 10 randomly timed check-ins during the 10-week intervention period
  Proportion of check-ins at which participant is carrying epinephrine auto-injector, measured using cell phone photographs

SECONDARY OUTCOMES:
Characterize adolescents' normative food allergy management practices | Year-long cohort study
  Characterize adolescents' normative food allergy management practices, measured comparing baseline and follow-up surveys that assess social challenges, out-of-home eating, allergen avoidance, and response to adverse events.
Characterize adolescents' normative food allergy management practices | Year-long cohort study
  Characterize adolescents' normative food allergy management practices, measured using periodic text-message questions that assess social challenges, out-of-home eating, allergen avoidance, and response to adverse events.
Develop a set of text message reminders to promote safer food allergy management among adolescents | 2-year project period
  Develop a set of text message reminders to promote safer food allergy management among adolescents by cognitively testing text message content

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Cannuscio, ScD, Principal Investigator — University of Pennsylvania; Jonathan Spergel, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupuis R, Spergel JM, Brown-Whitehorn TF, Troxel AB, Kenney EL, Block JP, Feuerstein-Simon R, Marti XL, Mollen CJ, Meisel ZF, Volpp KG, Gortmaker SL, Cannuscio CC. Incidence of food allergic reactions among adolescents engaged in food allergy management. Ann Allergy Asthma Immunol. 2025 Jun;134(6):719-723.e2. doi: 10.1016/j.anai.2025.02.023. Epub 2025 Mar 9. PMID 40068800